CLINICAL TRIAL: NCT01889251
Title: A Phase III Study of A01016 125μg Intravitreal Injection in Subjects With Symptomatic Vitreomacular Adhesion - Comparison Study to Sham Injection
Brief Title: A Phase III Study of A01016 in Subjects With Symptomatic Vitreomacular Adhesion
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: J-12-075
Record Dates: First submitted 2013-06-26; First posted 2013-06-28 (Estimated); Results first posted 2015-10-29 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Symptomatic Vitreomacular Adhesion
Keywords: Vitreomacular Adhesion; Vitreomacular Traction; Vitreomacular Traction Syndrome; Vitrectomy; Central Visual Field Defect; Blind Spot; Intravitreal Injection; Macula; Retina; Decreased Visual Acuity; Visual Complaint; SD-OCT; Macular Hole
MeSH Terms: conditions — Scotoma; Retinal Perforations | interventions — microplasmin; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ocriplasmin (Experimental): Ocriplasmin administered as a single intravitreal injection to the study eye at baseline
  Interventions: Drug: Ocriplasmin
- Sham injection (Sham Comparator): Single sham injection to the study eye at baseline
  Interventions: Drug: Sham injection

INTERVENTIONS:
Drug: Ocriplasmin
  Other Names: A01016
  Arms: Ocriplasmin
Drug: Sham injection
  Arms: Sham injection

SUMMARY:
The purpose of this study is to evaluate the superiority regarding vitreomacular adhesion (VMA) resolution of a single intravitreal injection of A01016 (Ocriplasmin) compared to sham-injection in subjects with symptomatic VMA.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic vitreomacular adhesion (VMA) which, in the opinion of the Investigator, is related to decreased visual function;
* Best corrected visual acuity (BCVA) of 20/25 or worse in the study eye;
* BCVA of 20/800 or better in the non-study eye;
* Provide written informed consent;
* Follow specified instructions during study period;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Evidence of proliferative retinopathy, exudative age-related macular degeneration, or retinal vein occlusion in the study eye;
* Vitreous hemorrhage or other opacification;
* High myopia in the study eye;
* Ocular surgery, laser photocoagulation treatment, or intravitreal injection(s) in the study eye in the prior 3 months;
* Uncontrolled glaucoma in the study eye;
* History of retinal detachment in either eye;
* Active infection in either eye;
* Pregnant or of child-bearing potential and not utilizing acceptable form of contraception;
* Participation in another investigational drug study within 30 days prior to this study;
* Other protocol-defined exclusion criteria may apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2013-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Group Manager, Clinical Development, Study Director — Alcon Japan, Ltd.
Locations (1):
- Contact Alcon for Trial Locations, Tokyo, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 40 study centers located in Japan.
Pre-assignment Details: Of the 251 enrolled, 79 subjects were exited as screen failures prior to randomization. This reporting group includes all randomized subjects (172).
Groups:
- Ocriplasmin: Single intravitreal injection to the study eye at baseline
Period: Overall Study
Arm/Group | Ocriplasmin | Sham Injection
Started | 115 | 57
Completed | 114 | 57
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized subjects, as randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ocriplasmin | Sham Injection | Total
Number analyzed (Participants) | 115 | 57 | 172
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.1 (7.3) | 68.6 (9.2) | 68.2 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 32 | 91
  Male | 56 | 25 | 81

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With Non-Surgical Resolution of Vitreomacular Adhesion (VMA)
Description: VMA (adhesion of the vitreous gel to the retina in an abnormally strong manner) was determined by masked Central Reading Center (CRC) Spectral Domain Optical Coherence Tomography (SD-OCT) evaluation. Only one eye (study eye) was analyzed. Proportion of subjects is reported as a percentage.
Time Frame: Day 28
Population: This analysis population includes all subjects who received study medication, completed at least 1 on-therapy study visit and had symptomatic VMA at baseline, as randomized, based on an intent to treat approach.
Measure: Number; unit: percentage of subjects
Arm/Group | Ocriplasmin | Sham Injection
Number analyzed (Participants) | 115 | 57
percentage of subjects | 52.2 | 1.8

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study (1 year, 2 months). This analysis group includes all subjects who received study medication, as treated. Note: One subject randomized to Ocriplasmin was inadvertently treated with Sham.
Description: An AE was defined as any untoward medical occurrence in a subject who is administered a study treatment regardless of whether or not the event has a causal relationship with the treatment. Ocular adverse events are presented for both study eye and non-study eye.
Arm/Group | Ocriplasmin | Sham Injection
Serious Adverse Events (participants affected / at risk) | 23/114 | 4/58
Other Adverse Events (participants affected / at risk) | 63/114 | 19/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ocriplasmin (N=114) | Sham Injection (N=58)
Macular hole (Eye disorders) | 11 | 3
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Vitreous adhesions (Eye disorders) | 2 | 1
Pneumonia (Infections and infestations) | 2 | 0
Retinal detachment (Eye disorders) | 3 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Ocular hypertension (Eye disorders) | 1 | 0
Angle closure glaucoma (Eye disorders) | 1 | 0
Intraocular pressure increased (Investigations) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Macular pseudohole (Eye disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ocriplasmin (N=114) | Sham Injection (N=58)
Conjunctival haemorrhage (Eye disorders) | 22 | 5
Vitreous floaters (Eye disorders) | 14 | 2
Anterior chamber cell (Eye disorders) | 13 | 3
Eye pain (Eye disorders) | 13 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 4
Conjunctival hyperaemia (Eye disorders) | 9 | 0
Visual impairment (Eye disorders) | 8 | 1
Corneal disorder (Eye disorders) | 8 | 0
Punctate keratitis (Eye disorders) | 7 | 1
Retinal detachment (Eye disorders) | 7 | 0
Intraocular pressure increased (Investigations) | 7 | 4
Constipation (Gastrointestinal disorders) | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.